CLINICAL TRIAL: NCT02031081
Title: Prucalopride Versus Placebo in Gastroparesis: Randomized Placebo-controlled Crossover Trial
Brief Title: Prucalopride Versus Placebo in Gastroparesis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Janssen Inc. (Industry)
Responsible Party: Principal Investigator, Christopher Andrews, Associate Professor, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PruGP
Record Dates: First submitted 2014-01-05; First posted 2014-01-09 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Gastroparesis; Diabetes Mellitus
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Period 1 (Experimental): A randomized assignment of prucalopride or placebo for a period of 28 days, crossover design
  Interventions: Drug: Prucalopride; Drug: Placebo
- Treatment Period 2 (Experimental): A randomized assignment of either prucalopride or placebo for a period of 28 days, crossover design. Subjects who received active drug in Treatment Arm 1 will receive placebo and vice versa.
  Interventions: Drug: Prucalopride; Drug: Placebo

INTERVENTIONS:
Drug: Prucalopride — 2 X 2 mg tablets (encapsulated) by mouth once daily for 28 days
  Other Names: Resotran
Drug: Placebo — 2 X 100mg tablets (encapsulated) by mouth once daily for 28 days
  Other Names: Lactose Monohydrate

SUMMARY:
The incidence of gastroparesis has been increasing among Canadians. Symptoms of discomfort include early satiety, stomach pain, nausea and vomiting. In addition, because gastroparesis slows digestion, it can lead to malnutrition and make controlling blood sugar even more challenging for diabetics. Mild cases of gastroparesis can be helped with dietary and lifestyle modifications but treatments for more severe symptoms are limited. There are several drugs called pro-kinetics available in Canada though results vary among patients and these often cause significant side effects. Recently, a drug called Prucalopride was approved for use in Canada to treat constipation. It has pro-kinetic properties and has been shown to cause few side effects. The investigators propose to test prucalopride as a treatment for gastroparesis by recruiting 30 patients from the Calgary area who have gastroparesis. The investigators will test the effects of this treatment by alternating 28 days of active treatment with prucalopride with 28 days of treatment with a non active placebo adding a two week break in between treatments. The order of the treatment will be randomized and neither the patients nor the investigators will know whether they are receiving the active treatment or the placebo until the study has been completely finished. The investigators will measure the effects using questionnaires that assess patient symptoms such as nausea and pain as well as quality of life during two gastric emptying tests and throughout the treatment periods. The effectiveness of the active treatment will be evaluated by comparing the extent of the change in symptoms before and after treatments and the difference in gastric emptying times as compared to the placebo treatment. The investigators will also monitor and track all possible side effects that patients experience during the study.

Study Hypotheses

In patients with gastroparesis:

1. Prucalopride 4 mg daily improves meal-related symptoms compared to placebo as defined by the change in cumulative meal-related symptoms. (primary endpoint).
2. Prucalopride 4 mg daily accelerates gastric emptying rate compared to placebo. (secondary endpoint).
3. A correlation exists between the effect of prucalopride on gastric emptying rate and symptom improvement.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-64 years
* Existing clinical diagnosis of gastroparesis for at least one year as judged by the study gastroenterologist based on past medical history, clinical symptoms
* Sufficiently symptomatic at time of proposed study (Minimum baseline postprandial satiety/fullness subscale of the Gastroparesis Cardinal Symptoms Index (GCSI) score of 1.5 or higher)
* Delayed gastric emptying (>10% retention at 4 hours) on standard solid meal scintigraphic emptying study within the previous year
* Normal upper endoscopy (with the exception of small bezoars) since the onset of symptoms
* If female of childbearing potential, a negative urine pregnancy test administered between consent and screening appointments
* Able to provide written informed consent

Exclusion Criteria:

* Clinical evidence (including physical exam and/or ECG) of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric or other disease that may interfere with the objectives of the study and/or pose safety concerns, including pregnancy or breastfeeding.
* Study entry ECG showing second or third degree heart block, left bundle branch block (LBBB) or acute ischemic changes
* Blood electrolytes (Na, K, CL) measured within past 6 months outside of normal reference ranges (except during an acute gastroparesis flare-up)
* Use of narcotics or promotility agents which cannot be stopped prior to study entry.
* Use of tricyclic antidepressants (at doses exceeding 25 mg/day) and/or macrolide antibiotics. (Stable doses of SSRI/SNRI antidepressants and/or non-macrolide antibiotics are permitted)
* Laxative use that cannot be stopped prior to the start of the study
* Participated in clinical trial with motility agents within past 30 days
* History of gastrointestinal surgery excepting appendectomy and/or cholecystectomy in the past, or any other major surgeries within 3 months
* Estimated GFR<30 measured within past 6 months.
* History of cardiovascular disorder including myocardial infarction, pacemaker or implanted defibrillator, or history of life-threatening arrhythmia

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-03; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change In Cumulative Meal-related Symptoms | Pre-intervention and on Day 28 for each of the two treatment periods
  Self assessment of 6 gastric related symptoms using a scale of 0-3 measured before and every 15 minutes during scintigraphic gastric emptying test.

SECONDARY OUTCOMES:
Gastric Emptying Rate | On Day 28 for each of the two treatment phases
  Percent remaining at 1, 2 and 4 hours will be determined from data gathered during 4 hour scintigraphic gastric emptying test

CONTACTS AND LOCATIONS:
Overall Officials: Christopher N Andrews, MD, MSc, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No